CLINICAL TRIAL: NCT06386653
Title: SPECT Imaging of EpCAM Receptors Using [123I]I-DARPIN-Ec1 in Lung and Ovarian Cancers Patients
Brief Title: Molecular Imaging of EpCAM Receptors Using [123I]I-DARPIN-Ec1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other); The Shemyakin and Ovchinnikov Institute of Bioorganic Chemistry (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: [123I]I-DARPIN-Ec1
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Ovarian Cancer
Keywords: Lung cancer; Оvarian cancer; [123I]I-DARPIN-Ec1; SPECT
MeSH Terms: conditions — Lung Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body planar scintigraphy and SPECT with [123I]I-DARPIN-Ec1 in lung cancer (Experimental): At least five (5) evaluable subjects with lung cancer.
  Interventions: Drug: Diagnostic injection of [123I]I-DARPIN-Ec1; Diagnostic Test: Whole-body planar scintigraphy with [123I]I-DARPIN-Ec1; Diagnostic Test: Whole-body SPECT with [123I]I-DARPIN-Ec1
- Whole-body planar scintigraphy and SPECT with [123I]I-DARPIN-Ec1 in ovarian cancer (Experimental): At least five (5) evaluable subjects with ovarian cancer.
  Interventions: Drug: Diagnostic injection of [123I]I-DARPIN-Ec1; Diagnostic Test: Whole-body planar scintigraphy with [123I]I-DARPIN-Ec1; Diagnostic Test: Whole-body SPECT with [123I]I-DARPIN-Ec1

INTERVENTIONS:
Drug: Diagnostic injection of [123I]I-DARPIN-Ec1 — A single intravenous injection of [123I]I-DARPIN-Ec1
  Other Names: [123I]I-DARPIN-Ec1 injection
Diagnostic Test: Whole-body planar scintigraphy with [123I]I-DARPIN-Ec1 — Gamma camera-based whole-body planar scintigraphy imaging 2, 4, 6, and 24 hours after a single intravenous injection of [123I]I-DARPIN-Ec1
  Other Names: [123I]I-DARPIN-Ec1 scintigraphy
Diagnostic Test: Whole-body SPECT with [123I]I-DARPIN-Ec1 — Whole-body SPECT at 2, 4, and 6 hours after a single intravenous injection of [123I]I-DARPIN-Ec1
  Other Names: [123I]I-DARPIN-Ec1 SPECT

SUMMARY:
The study should evaluate the biological distribution of [123I]I-DARPIN-Ec1 in patients with lung and ovarian cancer

The primary objective are:

1. To assess the distribution of [123I]I-DARPIN-Ec1 in normal tissues and tumors at different time intervals.
2. To evaluate dosimetry of [123I]I-DARPIN-Ec1.
3. To study the safety and tolerability of the drug [123I]I-DARPIN-Ec1 after a single injection in a diagnostic dosage.

The secondary objective are:

1. To compare the obtained [123I]I-DARPIN-Ec1 SPECT imaging results with the data of CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) studies in lung and ovarian cancer patients.

DETAILED DESCRIPTION:
The overall goal is to study the effectiveness of SPECT imaging lung and ovarian cancer using [123I]I-DARPIN-Ec1.

Phase I of the study:

Biodistribution of [123I]I-DARPIN-Ec1 in patients with lung and ovarian cancer .

The main objectives of the study:

1. To evaluate the distribution of [123I]I-DARPIN-Ec1 in normal tissues and tumors in patients with lung and ovarian cancer at different time intervals.
2. To evaluate dosimetry of [123I]I-DARPIN-Ec1 based on the pharmacokinetic parameters of the drug after a single intravenous administration.
3. To study the safety of use and tolerability of the drug [123I]I-DARPIN-Ec1 after a single intravenous administration in a diagnostic dosage.

Additional research tasks:

1. To conduct a comparative analysis of the diagnostic information obtained in the visualization of lung and ovarian cancer by SPECT using [123I]I-DARPIN-Ec1 with data obtained by CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) research of postoperative material.

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labeled tracer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of lung and ovarian cancer with histological verification.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of lung and ovarian cancer with histological verification.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
* Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body [123I]I-DARPIN-Ec1 uptake value (%) | 24 hours
  Whole-body [123I]I-DARPIN-Ec1 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based [123I]I-DARPIN-Ec1 value in tumor lesions (counts) | 6 hours
  [123I]I-DARPIN-Ec1 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based [123I]I-DARPIN-Ec1 uptake value (counts) | 6 hours
  Focal uptake of [123I]I-DARPIN-Ec1 in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of [123I]I-DARPIN-Ec1 uptake coinciding with tumor lesions (counts) will be divided by the value of [123I]I-DARPIN-Ec1 uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Percent of cases with abnormal findings in physical examination, vital signs and ECG associated with [123I]I-DARPIN-Ec1 injections. | 24 hours
  The safety attributable to [123I]I-DARPIN-Ec1 injections will be evaluated based on the assessments of physical examination, vital signs and ECG (percent of cases with abnormal findings relative to baseline).
Percent of cases with abnormal laboratory test results associated with [123I]I-DARPIN-Ec1 injections associated with [123I]I-DARPIN-Ec1 injections. | 24 hours
  The safety attributable to [123I]I-DARPIN-Ec1 injections will be evaluated based on the blood and urine laboratory tests (percent of cases with abnormal findings relative to baseline)
Incidence and severity of adverse events associated with [123I]I-DARPIN-Ec1 injections | 24 hours
  The safety attributable to [123I]I-DARPIN-Ec1 injections will be evaluated based on the rate of adverse events (percent)
Percent of cases requiring administration of concomitant medication due to [123I]I-DARPIN-Ec1 injections | 24 hours
  The safety attributable to [123I]I-DARPIN-Ec1 injections will be evaluated based on the rate of administration of concomitant medication (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, Prof, Study Director — Oncology Research Institute of Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared on request after consideration of requester's application.
Supporting Information: Study Protocol, SAP
Time Frame: Three years after completions of the study.
Access Criteria: Review of requester's application submitted to the Principal Investigator.